CLINICAL TRIAL: NCT06083116
Title: Evaluation of Drug-drug Interaction Between Henagliflozin Proline and Hydrochlorothiazide in Healthy Chinese Volunteers
Brief Title: Drug-Drug Interaction Study Between Henagliflozin Proline and Hydrochlorothiazide
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR3824-118
Record Dates: First submitted 2023-10-06; First posted 2023-10-13 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Diabetes in Adults

STUDY DESIGN:
Intervention Model Description: Evaluation of drug-drug interaction between Henagliflozin Proline and Hydrochlorothiazide. A single-center, single-arm, open-label, multi-dose, three-period study was conducted in healthy Chinese volunteers.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- healthy subjects (Experimental)
  Interventions: Drug: Hydrochlorothiazide、Henagliflozin Proline

INTERVENTIONS:
Drug: Hydrochlorothiazide、Henagliflozin Proline — Hydrochlorothiazide and Henagliflozin Proline

SUMMARY:
A single-center, single-arm, open-label, multi-dose, three-period study was conducted in healthy Chinese volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male;
2. Age 18-40 (including threshold);
3. Weight ≥ 50 kg, body mass index (BMI): 19.0~26.0 kg/m2 (including critical value);
4. Volunteers (and their spouses) must not plan for childbearing or sperm donation within one month prior to signing the informed consent form and from the period of taking the research drug until three months after stopping it;
5. Be able to communicate well with the investigators and understand and comply with the requirements in this study.

Exclusion Criteria:

1. Those have allergic constitution, or those with a known history of allergies to study drug or their excipients
2. Physical examination, vital signs, blood-routine examination, blood biochemistry, infectious disease screening, coagulation function, urine-routine examination, chest x-ray, B ultrasound and other examination results are abnormal and judged by the research doctor as clinically significant.
3. Hepatitis B surface antigen positive, hepatitis C antibody positive, HIV antibody positive, syphilis antibody positive;
4. Previous history of urinary tract infection or genital infection;
5. Previous history of hypoglycemia and other important diseases;
6. Those who have used other experimental drugs or medical devices within 3 months before screening;
7. Those who seek medical within 3 months prior to screening, which are judged by the research doctor to be unfit for participants;Those who have undergone any surgery within 6 months prior to screening;
8. Those who donate blood or other reasons of bleeding cause the total loss of blood more than 400mL or receive blood transfusions within 3 months before screening;
9. Have used any drugs in two weeks prior to taking the study drug;
10. Can not comply with the unified dietary arrangement;
11. Alcohol abuse, or those who smoke more 5 cigarettes per day in the 6 months prior to screening;
12. Positive alcohol breath test,or positive drug screening;
13. From 3 days before taking the study drug, subjects have xanthine-rich beverages or food, or grapefruit and other fruits or juices that may affect metabolism;
14. Subjects who are judged by researchers to be unsuitable for participating in this test.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2019-08-28 (Actual); Primary Completion 2019-10-10 (Actual); Study Completion 2019-10-10 (Actual)

PRIMARY OUTCOMES:
Steady-state pharmacokinetics parameters of Henagliflozin Proline: AUCτ,ss | Day 10, Day 14
Steady-state pharmacokinetics parameters of Henagliflozin Proline: Css, max | Day 10, Day 14
Steady-state pharmacokinetics parameters of Hydrochlorothiazide: AUCτ,ss | Day 4, Day 14
Steady-state pharmacokinetics parameters of Hydrochlorothiazide: Css, max | Day 4, Day 14

SECONDARY OUTCOMES:
Pharmacokinetics parameters of Henagliflozin Proline: Tmax | Day 10, Day 14
Pharmacokinetics parameters of Henagliflozin Proline: t1/2 | Day 10, Day 14
Pharmacokinetics parameters of Henagliflozin Proline: CL/F | Day 10, Day 14
Pharmacokinetics parameters of Hydrochlorothiazide: Tmax | Day 4, Day 14
Pharmacokinetics parameters of Hydrochlorothiazide: t1/2 | Day 4, Day 14
Pharmacokinetics parameters of Hydrochlorothiazide: CL/F | Day 4, Day 14
Accumulated urine electrolyte excretion 24 hours after administration | Day 4, Day 14
Urinary volume at 24 hours after administration | Day 4, Day 10, Day 14
Accumulated urine glucose excretion within 24 hours after administration | Day 10, Day 14
Adverse events | Day 4, Day 14

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Xuhui Central Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chen Q, Yu C, Wu Q, Song R, Liu Y, Feng S, Yu C, Jia J. Evaluation of Drug-Drug Interaction Between Henagliflozin and Hydrochlorothiazide in Healthy Chinese Volunteers. Drug Des Devel Ther. 2024 May 29;18:1855-1864. doi: 10.2147/DDDT.S433377. eCollection 2024. PMID 38828023